CLINICAL TRIAL: NCT07183553
Title: The Effect Of Family-Centered Care Approach On Physiological Parameters And Follow-Up Tıme In Infants Receiving Hıgh-Flow Nasal Oxygen Therapy Wıth The Diagnosis Of Lower Respiratory Tract Infection
Brief Title: The Effect of a Family-Centered Care Approach on Infants Receiving High-Flow Nasal Oxygen Therapy
Status: Completed | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, RUMEYSA NUR YILMAZ, Nurse, Ankara Etlik City Hospital
Other Study IDs: HITU-SBF-RNY-01
Record Dates: First submitted 2025-07-09; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Lower Respiratory Tract Infection
Keywords: Family-centered care; high-flow nasal oxygen therapy; lower respiratory tract infection; respiratory failure; nursing; infant
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- intervention group: After completing the data in the first section of the Mother and Baby Introductory Information Form, which includes information about the mother and baby, and the Family-Centered Care Scale, the mothers received one-on-one information, which lasted approximately 30 minutes, based on the content of the prepared education booklet. The education booklet covered topics on family-centered care, clinical equipment, steam application, and postural drainage. The mother was supported by a nurse throughout the care process until discharge. Maternal care practices were implemented under the supervision of the nurse, and questions about care were answered. The Family-Centered Care Scale was administered before discharge.
  Interventions: Other: maintenance training
- control group: After completing the data in the first section of the Mother and Baby Information Form, which includes information about the mother and baby, and the Family-Centered Care Scale, the mothers were trained by the nurses in accordance with the standard training content of the service. This content included general service rules, general materials used in the service, and a service introduction. Families were also provided with basic information about high nasal flow, including what it means. Care practices were implemented by the nurse until discharge. The Family-Centered Care Scale was administered at discharge.

INTERVENTIONS:
Other: maintenance training — information has been provided in accordance with the content of the training booklet.
  Groups: intervention group

SUMMARY:
This research is an experimental study of randomized control with pre-test - post-test control group.

The aim of this study is to determine the effect of family-centered care approach on physiological parameters and follow-up time in infants with respiratory failure diagnosed with lower respiratory tract infection and receiving high-current oxygen therapy

DETAILED DESCRIPTION:
The population of the study consisted of babies and their mothers who were receiving high-flow nasal oxygen therapy in the baby wards of Ankara Etlik City Hospital between December 2024 and March 2025.After receiving written consents with the volunteer consent form from the mothers who agreed to participate in the study, the volunteers were divided into intervention and control groups using the "computerized randomization method" (www.randomizer.org ). Patients were distributed to two groups according to the randomization list and all groups were informed about how to fill out follow-up forms. In both groups, the data in the section on introductory characteristics of the mother and baby in the first part of the Mother and Baby Introductory Information Form were filled in. A pre-test was administered with the family-centered care scale. The data related to the measurements of life signs (body temperature, pulse, respiration, oxygen saturation and blood pressure) contained in the introductory characteristics section of the baby were obtained from the patient's file and recorded. The intervention group received the "Family-Centered Care Program" and the control group received the standard care program of the clinic.The families in the intervention group were given training and information about family-centered care and were given an educational booklet that had been prepared. Before discharge, a post-test was conducted on both groups using the family-centered care scale.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Literate,
* Agreeing to participate in the study,
* Oriented to person, place, and time,
* No visual (except for those with improved vision using visual aids) or auditory communication difficulties (except for those with improved hearing using hearing aids) that would prevent them from understanding and expressing the information provided,
* No speech impairments/communication problems,
* Mothers of infants aged 28 days to 2 years, receiving high-flow oxygen therapy due to a lower respiratory tract infection, and without any chronic disease.

Exclusion Criteria:

* Mothers who did not speak or read Turkish,
* who were participating in a different study conducted at the clinic, were not included in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study included babies and their mothers who were treated in baby wards and received high-flow nasal oxygen therapy.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Family Centred Care Scale | three days
  The Family-Centered Care Scale (FCCS), consists of two sections. Both sections contain the same questions. The scale, divided into two sections for importance and consistency, consists of seven items. Each item is scored from 1 to 5. The lowest possible score is 7, and the highest is 35. As the total score increases, satisfaction with family-centered care increases in direct proportion to the score obtained from the scale. The items consist of questions regarding the evaluation of the nursing care received by parents during their hospital stay. The importance section evaluates the level of care shown by the nurses, and the consistency section evaluates the level of care shown by the nurses in the child's care. In the scale's evaluation, the importance and consistency scores are added together to form a single score.

CONTACTS AND LOCATIONS:
Locations (1):
- Hitit University, Çorum, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided